CLINICAL TRIAL: NCT04410536
Title: Home-withdrawal Program Combined With Behavioural Approach in Patients With Medication Overuse Headache During Covid-19 Emergency: Incidence of Relapses in Overuse and Changes in Impact at One Year Follow up
Brief Title: Home Detox in Medication Overuse Headache (MOH) During Covid-19 Emergency
Acronym: MOHC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MOH
Record Dates: First submitted 2020-05-25; First posted 2020-06-01 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Migraine, Hemicrania
MeSH Terms: conditions — Migraine Disorders | interventions — Bridge Therapy

STUDY DESIGN:
Intervention Model Description: withdrawal program will be performed at home
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Symptomatic drugs - bridge theray - mindfu (Other): 1. abrupt withdrawal of overuse symptomatic drugs, with possibility to use indomethacin suppository 50-100 mg or an oral triptan, on maximum 3 days/10 days, only in case of very severe headache- and to use metoclopramide i.m. injection in case of vomiting;
  2. oral administration of a bridge therapy to reduce the withdrawal symptoms and rebound headache (prednisone 25 mg , 2 tablets after breakfast for 5 days, one tablet for 3 days, half tablet for 2 days ; bromazepam 1.5 mg, 1 tablet after breakfast, lunch and dinner for every day; pantoprazole 40 mg, 1 tablet after dinner every day);
  3. mindfulness practice daily with standard sessions by smartphone 6 minutes per day.
  Interventions: Drug: Symptomatic drugs; Drug: Bridge therapy; Behavioral: Mindfulness program

INTERVENTIONS:
Drug: Symptomatic drugs — indomethacin suppository 50-100 mg or an oral triptan, on maximum 3 days/10 days, only in case of very severe headache- and to use metoclopramide
Drug: Bridge therapy — prednisone 25 mg , 2 tablets after breakfast for 5 days, one tablet for 3 days, half tablet for 2 days ; bromazepam 1.5 mg, 1 tablet after breakfast, lunch and dinner for every day; pantoprazole 40 mg, 1 tablet after dinner every day
Behavioral: Mindfulness program — home based withdrawal program

SUMMARY:
Medication Overuse Headache (MOH) is a disabling condition that affects the 2% of migraine population. Medication overuse (MO) makes this condition very difficult to treat. The literature of the last decades confirm the efficacy of withdrawal for patients with medication overuse, but it is also confirmed that patients have to be carefully followed after withdrawal to avoid relapses and to improve the clinical benefit of the therapeutic approach. Clinical results can be improved when traditional therapies are combined with behavioral approaches in particular mindfulness, that help patient to become more conscious about their symptoms and able to manage pain without medication. As the emergency situation due to the Corona-virus pandemic phenomenon in Italy, the regular clinical practice adopted for patients with CM-MO has changed in the last weeks: patients cannot come to the hospital for the withdrawal iv therapy and for regular follow up as the reduced mobility due to the emergency in particular in the Lombardia region, but all over Italy. So the investigators propose a pilot study to enforce the application of a Home-program for the withdrawal procedure for patients and the use of technology like smartphone and video calls so that patients can continue to be followed in their therapeutic process by using behavioral support and mindfulness practice. Patients will perform the withdrawal program at home, by oral administration of therapies, with specific instructions and education. Also the information for behavioral approach and mindfulness practice will be given, to use every day at home. Daily standardized mindfulness sessions of 12 minutes on their smartphone will be combined with weekly video-call to evaluate the clinical condition and to encourage the use strategies for pain management. Face-to-face visits at the follow up every three months will be scheduled. This modality will allow the patients to continue their therapeutic process and to be regularly followed during the one year after withdrawal.

DETAILED DESCRIPTION:
Background and significance Medication Overuse Headache (MOH) is a disabling pain syndrome with a prevalence of 2% in the general population, and which affects patients suffering from primary headaches, mainly those with Chronic Migraine (CM). This condition is very difficult to treat. The literature of the last decades confirmed the need to stop overuse through withdrawal (or detoxification programs) as an essential step in the treatment strategy , and high rates of successful outcomes are reported by several studies and reviews, although not all patients receiving treatment are able to stop MO or to reduce significantly the frequency of headaches. Remission rates range from 60% to 83% in studies with a 1-year follow-up, with an average relapse rate into MOH of 32.8% in a review on several studies from different countries, which is similar to the relapse into CM of 21.5% and into MOH of 33.9% found in a sample from our group . Literature data showed that patients need to be carefully followed after withdrawal to avoid relapses in overuse and to improve the clinical benefit, adding anti-migraine prophylaxi . Furthermore, different clinical experiences confirmed the effectiveness of interventions based on out-patient withdrawal programs and education and support to the correct use of medications to patients, and published evidence - also from our research group - supports the role of standardized behavioural approaches . The aspect of feasibility of these treatments is not regularly reported in published studies, but it can be estimated that a proportion of patients discontinue the treatment protocols, with a drop-out rate around 15-20% at one year from withdrawal., as it was 11% after 6 months, and 18% after 1 year in the seminal study by Katsarawa et al, and 9% after one year from withdrawal in a previous study from our research group . According to our protocols at the Headache Center, the withdrawal program is performed at hospital, either in an in-patient setting or in day-hospital setting. This program includes abrupt interruption of the overused drugs, intravenous therapy, educational support, rescue treatments for severe headaches, and prescription of a specific pharmacological prophylaxis for migraine prevention. Furthermore, standardized behavioural therapies are used during the treatment period, and during the follow up, particularly by approaches based on mindfulness practice - which usually delivered in groups of 4 - 8 patients . This approach may be particularly useful in helping patients to obtain a better outcome. All the above discussed considerations are even more relevant in this emergency situation due to the Corona-virus pandemic phenomenon in Italy, with its consequences on mobility of patients and clinical practice. In order to promote different modalities to respond to the needs of patients suffering from this disabling condition during the emergency, exercise-based telemedicine and smartphone applications seem very appropriate, as they have been recently tested in the management of chronic pain conditions . This preliminary study will be performed considering that the Covid-19 emergency reduced significantly our possibility to hospitalize patients for withdrawal treatments as well as the mobility of patients, particularly those living in other Italian regions than Lombardy, and in view of providing an effective and somewhat innovative treatment program for MOH and CM patients. The proposed treatment intervention is based on our experience, and on published reports, but it specifically includes a home based withdrawal program, several visits performed as Video calls, and educational and support strategies aimed to develop skills to reduce overuse and to cope with pain by a standardized behavioural approach based on mindfulness - which will be delivered mainly by telemedicine and smartphone applications. The aim of this pilot study is to assess the feasibility and the effectiveness at long-term on relevant outcomes of a specific protocol, designed to be appropriate during the emergency situation due to COVID-19 epidemic, by an approach that is alternative to current practice, particularly as far as avoiding the need for hospitalization, reducing face-to-face hospital visits taking advantage of facilities offered by new technologies, besides including innovative and emerging treatment choices, namely a behavioural approach base on mindfulness.

ELIGIBILITY:
Inclusion Criteria:

age >18 yrs diagnosis of MOH and CM (1) written informed consent

Exclusion Criteria:

co-existent severe medical or psychiatric illnesses, documented by specific previous diagnoses seizures use of opioids

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Drop out rates | at 12 months
  Drop-out rates after withdrawal treatment

SECONDARY OUTCOMES:
Absence of Medication Overuse Headache (MOH) | at 12 months from withdrawal program (assessed by Daily Diary Card)
  Percentages of patients with absence of Medication Overuse Headache

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Istituto Neurologico C. Besta, Neuroalgology Unit, Milan, Milano, Italy

IPD SHARING:
Plan to Share IPD: No